CLINICAL TRIAL: NCT02741440
Title: Natural History of Spinocerebellar Ataxia Type 7 (SCA7)
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160090; 16-EI-0090
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12-02

CONDITIONS: Spinocerebellar Ataxia
Keywords: Spinocerebellar Ataxia; Natural History
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected Participants: Twenty-five (25) participants with molecularly-confirmed SCA7

SUMMARY:
Background:

Spinocerebellar ataxia type 7 (SCA7) is a disease in which people have problems with coordination, balance, speech and vision. It is caused by a change in the ATXN7 gene. A mutation in this ATXN7 gene causes changes in eye cells, which can lead to vision loss. There is no cure for SCA7 but researchers are looking for possible treatments. Researchers need more information about SCA7. They want to collect vision and neurology related data from people with SCA7. They want to learn how and what changes in the eye and brain when the ATXN7 gene isn t working properly.

Objective:

To learn more about SCA7 and its progression.

Eligibility:

People ages 12 and older with SCA7.

Design:

Participants will be screened with medical history and genetic testing from a previous National Eye Institute study or their personal physician.

Participants will have at least 7 visits over 5 years. They will have 2 visits during the first week of the study. Then they will be asked to come back every year for the next 5 years. Each visit will last several days and will include:

* Medical and eye history
* Several eye tests: some will include dilating the pupil with eye drops and taking photos or scans of the eyes.
* Electroretinography (ERG): Participants will sit in the dark with their eyes patched for 30 minutes. After this, the patches will be removed and contact lenses put into the eyes. They will watch flashing lights and information will be recorded.
* Neurological exams: Sensation, strength, coordination, reflexes, attention, memory, language, and other cognitive functions will be tested.
* Brain MRI: They will lie in a machine that takes pictures of the brain.
* Blood and urine tests
* Optional skin biopsy: About 3 millimeters of skin will be removed for more research testing; this is half the size of a pencil eraser.

DETAILED DESCRIPTION:
Objective:

Spinocerebellar Ataxia, type 7 (SCA7) is an autosomal dominant neurodegenerative disease characterized by progressive ataxia, retinal degeneration, and marked genetic anticipation. The objectives of this study are to 1) establish a cohort of participants with molecularly-confirmed SCA7 in anticipation of future clinical trials, 2) create a repository of plasma, DNA, and skin fibroblast samples from the accrued cohort of SCA7 participants, 3) formulate clinical outcome measures for future studies, and 4) acquire and perform preliminary analyses of data that may advance our understanding of the progression of retinal and neurodegeneration associated with molecularly-confirmed SCA7.

Study Population:

Twenty-five (25) participants, ages 12 and above, with molecularly-confirmed SCA7 will be accrued for this study.

Design:

In this natural history study, participants will be followed for at least five years. Because three years may be required to enroll 25 participants, this study will last at least eight years. All participants will undergo a standardized medical/ophthalmic history and a complete baseline eye examination, including non-invasive electrophysiology (e.g., electroretinography), psychophysiology (e.g., microperimetry, static perimetry), and diagnostic imaging examinations (e.g., optical coherence tomography). In addition, participants will undergo a detailed neurology exam, neuroimaging (MRI, including special sequences) and consult with speech pathology and/or other rehabilitation services, audiology, and neuropsychology.

To establish baseline, the participants will undergo two separate detailed eye examinations and a single neurology/neuroimaging examination within a one to two week period. Afterwards, they will return to the NEI clinic annually until the last-enrolled participant has completed a minimum of five study visits. Follow-up visits will consist of a single detailed eye exam, a single detailed neurology/neuroimaging exam, and follow-up with appropriate consultants. Participants may be seen at more frequent intervals at the investigators discretion, depending on the clinical and research situation. Participants will be required to submit a blood sample for research, and they will have the option to provide a skin biopsy to facilitate research at a cellular level.

Outcome Measures:

The primary outcome for this study is determination of the amplitude and time of photopic and scotopic responses on electroretinogram. Secondary outcomes include changes in visual acuity, microperimetry, peripheral visual field, color vision, macular thickness, and neurologic outcome variables. Exploratory outcomes for this study include: 1) the formulation of clinical outcome measures for future studies and 2) the acquisition and preliminary analysis of data that may advance our understanding of the progression of retinal and neurodegeneration associated with molecularly-confirmed SCA7. Cells from skin biopsies may be grown in the laboratory to better understand SCA7, including the evaluation of potential treatments.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant must be 12 years of age or older.
2. Participant must be able to understand and sign the protocol s informed consent document on their own behalf OR, in the case of a minor, have a legal guardian/parent with the ability to do the same.
3. Participant must be able to produce a recordable electroretinogram (ERG).
4. Participant must have the ability to cooperate the required testing. Participants unable to cooperate with one or more tests may be included only at the discretion of the Principal Investigator.
5. Participant must be willing and able to provide a blood sample.
6. Any female participant of childbearing potential must agree to have pregnancy testing prior to undergoing MRI.
7. Participant has molecularly-confirmed, symptomatic SCA7, as defined by CAG repeat expansion in the ATXN7 gene of greater than 35 repeats. Accrual will be biased towards those with lower numbers of abnormal repeats (above 35 repeats) as they are most likely to be able to cooperate with testing. Participants who have clinical findings consistent with SCA7 and a relative who has had molecular diagnosis, may be included in the study with subsequent confirmation of the number of repeats. Patients who have clinical findings consistent with SCA7, but no molecular diagnosis may be evaluated under an NEI screening, genetics bank, or evaluation and treatment protocol with subsequent molecular diagnosis performed within six months of their initial visit.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Participant is unable to cooperate with ophthalmic/neurologic testing, including inability to undergo brain MRI without sedation.
2. Participant has comorbidity, unrelated to ocular pathology, compromising the ability to view/image the retina and/or record an ERG.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from neurology, genetics, and ophthalmology practices across the nation, as well as from the SCA7 patient support group (e.g., The National Ataxia Foundation). All advertisements will undergo IRB-approval before release. Referrals from investigators for participants under the 08-EI-0102 or 15-EI-0128 NEI protocols may be accepted.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2016-07-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude and time of photopic and scotopic responses on electroretinogram | Baseline to Years 1-5
  Determine the amplitude and time of photopic and scotopic responses on electroretinogram

SECONDARY OUTCOMES:
changes in visual acuity, microperimetry, color vision, macular thickness, neurologic (including neuroimaging) outcome variables, eye movement recordings (e.g., saccadic velocity) and results of neuropsychologic testing | Baseline to years 1-5
  changes in visual acuity, microperimetry, color vision, macular thickness, neurologic (including neuroimaging) outcome variables, eye movement recordings (e.g., saccadic velocity) and results of neuropsychologic testing

CONTACTS AND LOCATIONS:
Overall Officials: Laryssa A Huryn, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-EI-0090.html